CLINICAL TRIAL: NCT01157247
Title: Intravenous Fentanyl or Local Anesthetic Infiltration for Pain Reducing During Spinal Needle Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croatian Society of Regional Anesthesia and Analgesia (Other)
Purpose: Treatment
Other Study IDs: CSRAA-CMA:007/03
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-06

CONDITIONS: Anesthesia; Spinal Puncture
Keywords: Anesthetic techniques; regional, spinal; Pain; lumbar puncture; Analgesia, local; Analgesia, intravenous
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group SNI (Other): Insertion of spinal needle with introducer
  Interventions: Procedure: Comparison of intravenous fentanyl and local anesthetic infiltration in pain reducing during spinal needle puncture
- Group SNI+LA (Other): Local infiltration of lidocaine was applied three minutes after insertion of spinal needle with introducer
  Interventions: Procedure: Comparison of intravenous fentanyl and local anesthetic infiltration in pain reducing during spinal needle puncture
- Group SNI+F (Other): Intravenous fentanyl was applied 3 min before insertion of spinal needle with introducer
  Interventions: Procedure: Comparison of intravenous fentanyl and local anesthetic infiltration in pain reducing during spinal needle puncture
- Group SN (Other): Spinal puncture was performed only with spinal needle without introducer, local anesthetic infiltration or intravenous fentanyl before spinal puncture.
  Interventions: Procedure: Comparison of intravenous fentanyl and local anesthetic infiltration in pain reducing during spinal needle puncture

INTERVENTIONS:
Procedure: Comparison of intravenous fentanyl and local anesthetic infiltration in pain reducing during spinal needle puncture

SUMMARY:
Background and Objectives: Spinal puncture is painful procedure which may cause patient refusal of spinal anesthesia in future surgery. It could be minimized with topical and infiltration local anesthetic or intravenous opioid application before procedure. Objective was efficacy of intravenous fentanyl in alleviating pain during spinal needle insertion.

Methods: Prospective, randomized study included 88 adults (33-55 ages, ASA I/II), scheduled for lower leg surgery. Patients were divided in four equal study groups: spinal needle (Quincke, 26G) with introducer (20G) was inserted alone, three minutes after local anesthetic infiltration (2 ml of 2% lidocaine, 25Gx11/4" needle) or intravenous fentanyl application (0.001 mg kg-1) and without local anesthetic, fentanyl and introducer. Pain was assessed immediately after procedure by VAS score. MAP, HR and SaO2 were recorded. Sedation was assessed by Ramsay score. Statistical analysis was performed by SPSS 11.0.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* ASA I or II status
* Scheduled for trauma or orthopedic surgeries of lower leg in spinal anesthesia

Exclusion Criteria:

* Patients with scoliosis
* Degenerative spine deformity
* A history of back surgery or back pain
* Pregnancy
* Perence of coagulopathy
* Systemic or local infection
* Allergy to amide-local anesthetics
* Neurologic damages and mental disability
* More than one spinal puncture attempt
* Patient who was unable to estimate pain score
* High Ramsay sedation score

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Traumatology, Zagreb, Croatia

REFERENCES:
- [Result] Almeida GP, Boos GL, Alencar TG, Oliveira Filho GR. [Onset of 1% lidocaine for skin infiltrative anesthesia]. Rev Bras Anestesiol. 2005 Jun;55(3):284-8. doi: 10.1590/s0034-70942005000300005. Portuguese. PMID 19471833
- [Result] Kaur G, Gupta P, Kumar A. A randomized trial of eutectic mixture of local anesthetics during lumbar puncture in newborns. Arch Pediatr Adolesc Med. 2003 Nov;157(11):1065-70. doi: 10.1001/archpedi.157.11.1065. PMID 14609894
- [Result] Calderon E, Pernia A, Roman MD, Perez AC, Torres LM. [Analgesia and sedation in the subarachnoid anesthesia technique: comparative study between remifentanil and fentanyl/midazolam]. Rev Esp Anestesiol Reanim. 2003 Mar;50(3):121-5. Spanish. PMID 12708207